CLINICAL TRIAL: NCT00078325
Title: A 12 Week, Randomized, Double Blind, Placebo Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of CEP 10953 (150 and 250 mg/Day) as Treatment for Adults With Residual Excessive Sleepiness Associated With Obstructive Sleep Apnea/Hypopnea Syndrome
Brief Title: Armodafinil (CEP-10953) in Treatment of Excessive Sleepiness Associated With Obstructive Sleep Apnea/Hypopnea Syndrome(OSAHS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C10953/3021/AP/MN
Record Dates: First submitted 2004-02-23; First posted 2004-02-25 (Estimated); Results first posted 2010-07-29 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Obstructive Sleep Apnea; Hypopnea
Keywords: Excessive Sleepiness; Obstructive Sleep Apnea; Obstructive Sleep Hypopnea; nCPAP; Cephalon; Cephalon, Inc; NUVIGIL
MeSH Terms: conditions — Sleep Apnea, Obstructive; Disorders of Excessive Somnolence | interventions — Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Armodafinil 250 mg/day
  Interventions: Drug: Armodafinil 250 mg/day
- 2 (Experimental): Armodafinil 150 mg/day
  Interventions: Drug: Armodafinil 150 mg/day
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Armodafinil 250 mg/day — Armodafinil 250 mg once daily in the morning
  Other Names: NUVIGIL; CEP-10953
  Arms: 1
Drug: Armodafinil 150 mg/day — Armodafinil 150 mg once daily in the morning
  Other Names: NUVIGIL; CEP-10953
  Arms: 2
Drug: Placebo — Matching placebo tablets once daily in the morning
  Arms: 3

SUMMARY:
The primary objective of this study is to determine whether treatment with Armodafinil (CEP-10953) is more effective than placebo treatment for patients with excessive sleepiness associated with obstructive sleep apnea/hypopnea syndrome (OSAHS) by measuring mean sleep latency from the Maintenance of Wakefulness Test (MWT) (30-minute version) (average of 4 naps at 0900, 1100, 1300, and 1500) and by Clinical Global Impression of Change (CGI-C) ratings (as related to general condition) at week 12, or last post-baseline visit.

ELIGIBILITY:
Inclusion Criteria:

Patients are included in the study if all of the following criteria are met:

1. Written informed consent is obtained.
2. The patient is an outpatient, man or woman of any ethnic origin, 18 to 65 years of age (inclusive).
3. The patient has a complaint of excessive sleepiness despite nCPAP therapy being effective and being a regular user of nCPAP therapy.
4. The patient has a current diagnosis of OSAHS according to International Classification of Sleep Disorders (ICSD) criteria.
5. The patient meets the following nCPAP therapy requirements:

   * Adequate education and intervention efforts to encourage nCPAP therapy use must be documented.
   * A patient's nCPAP therapy regimen must be stable for at least 4 weeks.
   * nCPAP therapy is shown to be effective, with effectiveness defined as having an apnea-hypopnea index (AHI) of 10 or less during nocturnal PSG, and, in the opinion of the investigator, nCPAP is effective therapy.
   * Following demonstration of effectiveness, evidence of regular nCPAP usage must be shown during a 2-week evaluation period (ie, nCPAP usage for at least 4 hours/night on at least 70% of the nights).
6. The patient is in good health as determined by a medical and psychiatric history, physical examination, ECG, and serum chemistry and hematology.
7. Women must be surgically sterile, 2 years postmenopausal, or, if of child-bearing potential, using a medically accepted method of birth control (ie, barrier method with spermicide, steroidal contraceptive [oral, implanted, and Depo-Provera contraceptives must be used in conjunction with a barrier method], or intrauterine device [IUD]) and agree to continued use of this method for the duration of the study.
8. The patient has a Clinical Global Impression of Severity of Illness (CGI-S) rating of 4 or more.
9. The patient has an ESS score of 10 or more.
10. The patient does not have any medical or psychiatric disorders that could account for the excessive sleepiness.
11. The patient is able to complete self rating scales and computer-based testing.
12. The patient is willing and able to comply with study restrictions and to attend regularly scheduled clinic visits as specified in this protocol.

Exclusion Criteria:

Patients are excluded from participating in this study if 1 or more of the following criteria are met:

1. has any clinically significant, uncontrolled medical or psychiatric conditions (treated or untreated)
2. has a probable diagnosis of a current sleep disorder other than OSAHS
3. consumes caffeine including coffee, tea and/or other caffeine containing beverages or food averaging more than 600 mg of caffeine per day
4. used any prescription drugs disallowed by the protocol or clinically significant use of over the-counter (OTC) drugs within 7 days before the second screening visit
5. has a history of alcohol, narcotic, or any other drug abuse as defined by the Diagnostic and Statistical Manual of Mental Disorders of the American Psychiatric Association, 4th Edition (DSM IV)
6. has a positive urine drug screen (UDS)
7. has a clinically significant deviation from normal in the physical examination
8. is a pregnant or lactating woman. (Any woman becoming pregnant during the study will be withdrawn from the study.)
9. has used an investigational drug within 1 month before the initial screening visit
10. has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery)
11. has a known clinically significant drug sensitivity to stimulants or modafinil

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2004-02; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 37 centers in the US and Canada. First patient enrolled: 19 February 2004/ Last patient last visit: 6 November 2004
Pre-assignment Details: 3 female patients withdrew after randomization but prior to receiving study drug (1 had a protocol violation and 2 were lost to follow-up)
Groups:
- Placebo: Matching placebo tablets once daily
Period: Overall Study
Arm/Group | Armodafinil 250 mg/Day | Armodafinil 150 mg/Day | Placebo
Started | 131 | 133 | 131
Completed | 110 | 114 | 120
Not Completed | 21 | 19 | 11
Not completed — Adverse Event | 15 | 10 | 5
Not completed — Protocol Violation | 2 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 5 | 3
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Physician Decision | 2 | 0 | 1
Not completed — Miscellaneous | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Armodafinil 250 mg/Day | Armodafinil 150 mg/Day | Placebo | Total
Number analyzed (Participants) | 131 | 131 | 130 | 392
Age, Categorical [Count of Participants; unit: Participants] — 3 female patients withdrew after randomization but prior to receiving study drug (1 had a protocol violation and 2 were lost to follow-up)
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 130 | 131 | 129 | 390
    >=65 years | 1 | 0 | 1 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 49.1 (8.74) | 49.3 (9.17) | 50.1 (9.43) | 49.5 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants] — 3 female patients withdrew after randomization but prior to receiving study drug (1 had a protocol violation and 2 were lost to follow-up)
  Participants
    Female | 42 | 34 | 40 | 116
    Male | 89 | 97 | 90 | 276
Region of Enrollment [Number; unit: participants]
  United States | 117 | 119 | 117 | 353
  Canada | 14 | 14 | 14 | 42

OUTCOME MEASURES:

1. Primary Outcome: Maintenance of Wakefulness Test (MWT)
Description: The MWT is an objective assessment of sleepiness that measures the ability of a subject to remain awake. Long latencies to sleep are indicative of a patient's ability to remain awake. The primary variable was the 30 minute MWT (average of 4 naps at 0900, 1100, 1300, and 1500) assessed at the last postbaseline observation.
Time Frame: change from baseline at 12 weeks
Population: Safety Analysis set of 392 total patients: 3 patients withdrew after randomization but prior to receiving study drug (1 had a protocol violation and 2 were lost to follow-up)
  Full Analysis set of 365 total patients: 27 patients that had withdrawn from the study were non-evaluable for efficacy.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Armodafinil 250 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 121 | 120 | 124
Minutes | 2.2 (8.07) | 1.7 (6.49) | -1.7 (8.59)
Statistical Analysis 1: Comparison: Armodafinil 250 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0001, ANOVA; Treatment and country as factors
Statistical Analysis 2: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0008, ANOVA; Treatment and country as factors

2. Primary Outcome: Clinical Global Impression of Change (CGI-C)
Description: The CGI-C represents a subjective measure of the patient's global health (clinician's rating of disease severity as compared with a pretreatment evaluation as assessed by the CGI-S). The CGI-C scale (change from baseline)categories include:1=Very much improved; 2=Much improved; 3=Minimally improved; 4=No change; 5=Minimally worse; 6=Much worse; and 7=Very much worse. Severity of illness (CGI-S) was assessed at baseline includes categories: 1=Normal; 2=Borderline ill; 3=Mildly (Slightly) ill; 4=Moderately ill; 5=Markedly ill; 6=Severely ill; and 7=Among the most extremely ill patients.
Time Frame: change from baseline at 12 weeks
Population: Safety Analysis set of 392 total patients (ITT): 3 patients withdrew after randomization but prior to receiving study drug (1 had a protocol violation and 2 were lost to follow-up)
Measure: Number; unit: Participants
Arm/Group | Armodafinil 250 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 121 | 120 | 124
Participants | 121 | 120 | 124
Statistical Analysis 1: Comparison: Armodafinil 250 mg/Day vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted for country
Statistical Analysis 2: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted for country

ADVERSE EVENTS:
Arm/Group | Armodafinil 250 mg/Day | Armodafinil 150 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 1/131 | 3/131 | 0/130
Other Adverse Events (participants affected / at risk) | 52/131 | 32/131 | 19/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil 250 mg/Day (N=131) | Armodafinil 150 mg/Day (N=131) | Placebo (N=130)
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Affective disorder (Psychiatric disorders) | 0 | 1 | 0
Personality disorder (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil 250 mg/Day (N=131) | Armodafinil 150 mg/Day (N=131) | Placebo (N=130)
Nausea (Gastrointestinal disorders) | 13 | 3 | 6
Dry Mouth (Gastrointestinal disorders) | 10 | 1 | 0
Headache (Nervous system disorders) | 27 | 19 | 11
Dizziness (Nervous system disorders) | 8 | 5 | 2
Insomnia (Psychiatric disorders) | 9 | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days